CLINICAL TRIAL: NCT07127471
Title: A Multicenter Prospective Randomized Controlled Trial of Linked-Color Imaging for Detection of Clinically Significant Serrated Lesions in Computer-Aided Water Exchange Colonoscopy
Brief Title: Computer-Aided Water Exchange Colonoscopy With and Without Linked-Color Imaging for Detection of Clinically Significant Serrated Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Evergreen General Hospital, Taiwan (Other)
Collaborators: Centre hospitalier de l'Université de Montréal (CHUM) (Other); King Chulalongkorn Memorial Hospital (Other); Ospedale Valduce, Como (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: WEAID with LCI
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Sessile Colonic Polyp; Serrated Lesion; Sessile Serrated Lesion; Colon Adenomas

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water exchange with AI-assisted detection (Active Comparator): The study employs standard high-definition colonoscopy video processors with integrated CADe system (CAD-EYE, EW10-EC02, Fujifilm) The ELUXEO 7000 system (Fujifilm) will be used in this study. During the insertion phase of water exchange (WE) colonoscopy, the air pump will be turned off, and the colon will be irrigated with warm water, using a flushing pump. WE involves simultaneous infusion of distilled water to facilitate luminal expansion and suction of unclean water. Withdrawal will begin with the patient in the left lateral position. Consistent techniques, ensuring adequate luminal distention and comprehensive fold examination, will be used. The CADe device will be activated during the withdrawal phase of the procedures, and it will provide real-time output in the form of a bounding box whenever the CADe device identifies a suspected polyp. All participating endoscopists possess experience and expertise in CADe systems, ensuring readiness before study initiation.
  Interventions: Device: Water exchange with AI-assisted detection
- Water exchange with AI-assisted detection and LCI (Experimental): The study employs high-definition colonoscopy video processors with integrated CADe (CAD-EYE, EW10-EC02, Fujifilm) and LCI systems (Fujifilm).The ELUXEO 7000 system will be used . During the insertion phase of water exchange (WE) colonoscopy, the air pump will be turned off, and the colon will be irrigated with warm water, using a flushing pump. WE involves simultaneous infusion of distilled water to facilitate luminal expansion and suction of unclean water. Withdrawal will begin with the patient in the left lateral position. Consistent techniques, ensuring adequate luminal distention and comprehensive fold examination, will be used. The CADe and LCI devices will be activated during the withdrawal phase of the procedures, and it will provide real-time output in the form of a bounding box whenever the CADe device identifies a suspected polyp. All participating endoscopists possess experience and expertise in CADe and LCI systems, ensuring readiness before study initiation.
  Interventions: Device: Water exchange with AI-assisted detection and LCI

INTERVENTIONS:
Device: Water exchange with AI-assisted detection — The study employs standard high-definition colonoscopy video processors with integrated CADe system (CAD-EYE, EW10-EC02, Fujifilm) The ELUXEO 7000 system (Fujifilm) will be used in this study. During the insertion phase of water exchange (WE) colonoscopy, the air pump will be turned off, and the colon will be irrigated with warm water, using a flushing pump. WE involves simultaneous infusion of distilled water to facilitate luminal expansion and suction of unclean water. Withdrawal will begin with the patient in the left lateral position. Consistent techniques, ensuring adequate luminal distention and comprehensive fold examination, will be used. The CADe device will be activated during the withdrawal phase of the procedures, and it will provide real-time output in the form of a bounding box whenever the CADe device identifies a suspected polyp. All participating endoscopists possess experience and expertise in CADe systems, ensuring readiness before study initiation.
  Arms: Water exchange with AI-assisted detection
Device: Water exchange with AI-assisted detection and LCI — The study employs high-definition colonoscopy video processors with integrated CADe (CAD-EYE, EW10-EC02, Fujifilm) and LCI systems (Fujifilm).The ELUXEO 7000 system will be used . During the insertion phase of water exchange (WE) colonoscopy, the air pump will be turned off, and the colon will be irrigated with warm water, using a flushing pump. WE involves simultaneous infusion of distilled water to facilitate luminal expansion and suction of unclean water. Withdrawal will begin with the patient in the left lateral position. Consistent techniques, ensuring adequate luminal distention and comprehensive fold examination, will be used. The CADe and LCI devices will be activated during the withdrawal phase of the procedures, and it will provide real-time output in the form of a bounding box whenever the CADe device identifies a suspected polyp. All participating endoscopists possess experience and expertise in CADe and LCI systems, ensuring readiness before study initiation.
  Arms: Water exchange with AI-assisted detection and LCI

SUMMARY:
The goal of this clinical trial is to compare the detection rate of clinically significant serrated lesions (CSSL) in participants undergoing water exchange (WE) colonoscopy with artificial intelligence (AI)-based computer-aided detection (CADe) for screening, surveillance, diagnosis for symptoms, or referred owing to a positive fecal immunochemical test (FIT) or guaiac fecal occult blood test (gFOBT) result. There will be two arms in this study: WE with AI-assisted CADe (WEAID) control and WEAID plus linked-color imaging (LCI). The main question it aims to answer is whether the addition of LCI into WEAID colonoscopy increases CSSL detection rate. Both groups use water instead of air to insert the colonoscope into the cecum. The control method uses CADe to help detect colonic lesions. The study method uses a combination of CADe and LCI to detect lesions. Researchers will compare CSSL detection rate to see if the addition of LCI increases the detection of CSSL during CADe-assisted WE colonoscopy.

DETAILED DESCRIPTION:
This will be a multicenter, unblinded investigators, prospective randomized controlled trial (RCT). Randomization (1:1 to WEAID alone and WEAID plus LCI) will be based on computer generated random numbers placed inside opaque sealed envelopes. The envelope (in pre-arranged order) will be opened to reveal the code when the colonoscopist is ready to insert the endoscope to begin the examination. This will be a comparison of two different methods with two arms (WEAID, WEAID-LCI) to see which one is better at detecting CSSL.

Patient recruitment will be conducted at 4 hospitals: University of Montreal Medical Center (CHUM), Quebec, Canada; Evergreen General Hospital, Taoyuan, Taiwan; King Chulalongkorn Memorial Hospital, Bangkok, Thailand; and Ospedale Valduce, Como, Italy. The study period is expected to be 2 years (from August 2025 to July 2027).

Patients aged 40-80 y/o at average risk of colorectal cancer who are willing to participate will sign an informed consent before starting the colonoscopy procedure. Separate parallel randomization will be set up at each site, stratified by investigator and indication of colonoscopy (screening, surveillance, diagnostic, or positive FIT or gFOBT result). Mode of sedation will include no sedation, on-demand sedation, conscious sedation or full sedation with propofol. Randomization will be carried out by computer-generated sequences.

The study employs standard high-definition colonoscopy video processors with integrated CADe system (CAD-EYE, EW10-EC02, Fujifilm). The ELUXEO 7000 system (Fujifilm) will be used. The same endoscopist performs the insertion and withdrawal of colonoscopy. The colonoscope will be inserted with WE method, instead of air insufflation. WE involves simultaneous infusion of distilled water to facilitate luminal expansion and suction of unclean water.

Control Method: One arm of the study will include CADe as the control method. The CADe system will be activated during the withdrawal phase of the procedures, and it will provide real-time output in the form of a bounding box whenever the CADe device identifies a suspected polyp.

Study method: The other arm entails the addition of a commercially available image-enhanced LCI technique (Fujifilm) to the CADe system. LCI will be activated during the withdrawal phase to enhance visualization of the lesions.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 40-80 years scheduled for average-risk screening colonoscopy, post-polypectomy surveillance, diagnosis for gastrointestinal symptoms (including unexplained iron deficiency anemia and clinically significant diarrhea of unexplained origin), or referred for colonoscopy owing to a positive fecal immunochemical test (FIT) or guaiac fecal occult blood test (gFOBT) result.

Exclusion Criteria:

* familial adenomatous polyposis and hereditary non-polyposis CRC syndrome
* personal history of serrated polyposis syndrome
* personal history of CRC
* history of inflammatory bowel disease
* previous colonic resection
* overt gastrointestinal bleeding
* emergency colonoscopy or inpatients
* planned EMR or ESD of large polyps
* colon stricture or obstruction
* contraindications to colonoscopy (eg, acute diverticulitis or toxic megacolon)
* antithrombotic therapy precluding complete polyp resection
* American Society of Anesthesiology classification of physical status >3
* pregnant women or women planning pregnancy
* refusal to provide a written informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1090 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Clinically significant serrated lesion (CSSL) detection rate | One week (after the colonoscopy procedure, when pathology report is released)
  Percentage of patients who have 1 or more histologically confirmed CSSLs, including sessile serrated lesions, traditional serrated adenomas, hyperplastic polyps measuring ≥10 mm anywhere in the colon, or hyperplastic polyps measuring 6-9 mm in the proximal colon (cecum to splenic flexure).

SECONDARY OUTCOMES:
Sessile serrated lesion (SSL) detection rate | One week (after the colonoscopy procedure, when pathology report is released)
  Percentage of patients who have 1 or more histologically confirmed SSL with or without dysplasia.
Proximal serrated lesion detection rate | One week (after the colonoscopy procedure, when pathology report is released)
  Percentage of patients who have 1 or more histologically confirmed proximal serrated lesions, including sessile serrated lesion, translational serrated adenoma, and hyperplastic polyp. The proximal colon includes the cecum, ascending colon, hepatic flexure, transverse colon, and splenic flexure.
High-risk neoplasm detection rate | One week (after the colonoscopy procedure, when pathology report is released)
  Percentage of patients who have 1 or more histologically confirmed advanced adenoma, or ≥5 low-risk adenomas (defined as 1 to 2 tubular adenomas <10 mm with low-grade dysplasia), or any serrated lesions ≥10 mm or with dysplasia. Advanced adenomas are defined as those adenomas meeting at least one of the following criteria: (1) size ≥10 mm, (2) presence of 25% villous components, and (3) high-grade dysplasia.
Adenoma detection rate | One week (after the colonoscopy procedure, when pathology report is released)
  Percentage of patients who have 1 or more histologically confirmed conventional adenomas.
Adenoma per colonoscopy | One week (after the colonoscopy procedure, when pathology report is released)
  Total number of histologically confirmed adenomas divided by the total number of colonoscopies.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Liang Cheng, MD, Study Chair — Evergreen General Hospital, Taoyuan; Rungsun Rerknimitr, MD, Principal Investigator — Center of Excellence for Innovation and Endoscopy in Gastrointestinal Oncology, King Chulalongkorn Memorial Hospital; Daniel von Renteln, MD, Principal Investigator — Research, Gastroenterology Division, University of Montreal Medical Center (CHUM); Franco Radaelli, MD, Principal Investigator — Gastroenterology Unit, Ospedale Valduce
Locations (4):
- University of Montreal Medical Center (CHUM), Montreal, Quebec, Canada
- Ospedale Valduce, Como, Italy
- Evergreen General Hospital, Taoyuan District, Taiwan
- King Chulalongkorn Memorial Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anderson JC, Hisey W, Mackenzie TA, Robinson CM, Srivastava A, Meester RGS, Butterly LF. Clinically significant serrated polyp detection rates and risk for postcolonoscopy colorectal cancer: data from the New Hampshire Colonoscopy Registry. Gastrointest Endosc. 2022 Aug;96(2):310-317. doi: 10.1016/j.gie.2022.03.001. Epub 2022 Mar 8. PMID 35276209
- [Background] Anderson JC, Rex DK, Mackenzie TA, Hisey W, Robinson CM, Butterly LF. Higher Serrated Polyp Detection Rates Are Associated With Lower Risk of Postcolonoscopy Colorectal Cancer: Data From the New Hampshire Colonoscopy Registry. Am J Gastroenterol. 2023 Nov 1;118(11):1927-1930. doi: 10.14309/ajg.0000000000002403. Epub 2023 Jul 7. PMID 37417792